CLINICAL TRIAL: NCT00489398
Title: Comparison of CL Wear Between Epinastine Hydrochloride and Olopatadine Hydrochloride
Brief Title: Comparison of CL Wear Between Two Allergy Drops
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Protocol changes
Sponsor: Hom, Milton M., OD, FAAO (Individual)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Milton M. Hom, OD, FAAO., Milton M. Hom, OD, FAAO.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 5316
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — epinastine; Olopatadine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: epinastine HCL and olopatadine HCL

SUMMARY:
Comparison of two allergy drops for enhancing comfort and performance of contact lens wear

DETAILED DESCRIPTION:
Contact lens patients will instill allergy drops and subjective and objective tests will be performed

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 18 years old
* Mild to moderate dry eye symptoms
* Likely to complete all study visits and able to provide informed consent

Exclusion Criteria:

* Current use of topical cyclosporine
* Known contraindications to any study medication or ingredients
* Active ocular diseases or uncontrolled systemic disease (blepharitis patients that are actively being treated or disease that is uncontrollable)
* Ocular surgery within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-07; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Contact lens objective and subjective clinical performance testing | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Milton M Hom, OD FAAO, Study Director — Private Practice